CLINICAL TRIAL: NCT03851939
Title: The Efficacy of Transarterial Chemoinfusion (TAI) Combine Toripalimab in Advanced Hepatocellular Carcinoma (HCC): A Prospective, Single-armed, Stage II Clinical Trial
Brief Title: The Efficacy of Transarterial Chemoinfusion (TAI) Combine Toripalimab in Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-158-01
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Transarterial Chemoinfusion (TAI) Combine Toripalimab
  Interventions: Combination Product: Transarterial Chemoinfusion (TAI) Combine Toripalimab

INTERVENTIONS:
Combination Product: Transarterial Chemoinfusion (TAI) Combine Toripalimab — Transarterial Chemoinfusion (TAI) Combine Toripalimab

SUMMARY:
To evaluate the efficacy of TAI combine toripalimab in advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years;
* ECOG PS≤1;
* proven advanced hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria;
* not previous treated for tumor;
* cannot accepted hepatectomy;
* the lab test could meet:

  * neutrophil count≥2.0×109/L;
  * hemoglobin≥100g/L;
  * platelet count≥75×109/L;
  * serum albumin≥35g/L;
  * total bilirubin<2-times upper limit of normal;
  * ALT<3-times upper limit of normal;
  * AST<3-times upper limit of normal;
  * serum creatine<1.5-times upper limit of normal;
  * PT≤upper limit of normal plus 4 seconds;
  * INR≤2.2;
* sign up consent;

Exclusion Criteria:

* cannot tolerate TAI or toripalimab;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorrhage or cardiac/brain vascular events within 30 days;
* pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-02-26 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of progression, assessed up to 36 months
  progression-free survival
ORR | From date of randomization until the date of death, assessed up to 36 months
  objective response rate

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 36 months
  overall survival
DCR | From date of randomization until the date of death, assessed up to 36 months
  disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China